CLINICAL TRIAL: NCT05151588
Title: A Phase II Single-arm Study of Tazemetostat With Docetaxel, Cisplatin, and 5-fluorouracil as Preoperative Treatment for Locally Advanced Potentially Resectable SMARCB1 (INI-1)- Deficient Sinonasal Carcinoma
Brief Title: Induction Chemotherapy and Tazemetostat for Locally Advanced SMARCB1-deficient Sinonasal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Victor H.F. Lee (Other)
Responsible Party: Sponsor-Investigator, Dr. Victor H.F. Lee, Clinical Associate Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMART-PNS
Record Dates: First submitted 2021-11-27; First posted 2021-12-09 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Sinonasal Carcinoma
Keywords: Induction therapy; Chemotherapy; Surgery
MeSH Terms: interventions — Docetaxel; Cisplatin; Fluorouracil; tazemetostat; Surgical Procedures, Operative; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: Induction treatment with docetaxel, cisplatin, 5-FU and tazemetostat followed by surgery or radical chemoradiation and maintenance tazemetostat
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction therapy followed by surgery and postoperative therapy (Experimental): Induction chemotherapy with docetaxel 75mg/m2 on day 1, cisplatin 75mg/m2 on day 1, 5-FU 750mg from day 1 to day 5, given every 3 weeks for 3 cycles and tazemetostat 800mg twice daily orally for 3 cycles, followed by radical surgery or radical chemoradiation, and maintenance tazemetostat 800mg twice daily orally for 6 months
  Interventions: Drug: Docetaxel; Drug: Cis Platinum; Drug: 5-FU; Drug: Tazemetostat; Procedure: Surgery; Other: Chemoradiation

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75mg/m2 intravenous infusion on day 1 every 3 weeks for 3 cycles as induction therapy
  Other Names: Taxotere
Drug: Cis Platinum — Cisplatin 75mg/m2 intravenous infusion on day 1 every 3 weeks for 3 cycles as induction therapy
  Other Names: CDDP
Drug: 5-FU — 5-FU 750mg/m2 intravenous infusion from day 1 to day 5 every 3 weeks for 3 cycles as induction therapy
  Other Names: 5-fluorouracil
Drug: Tazemetostat — Tazemetostat 800mg twice per day orally in continuously for 3 cycles as induction therapy and maintenance therapy
  Other Names: TAZVERIK
Procedure: Surgery — Radical surgery
  Other Names: Resection
Other: Chemoradiation — Chemoradiation as either radical treatment or post-operative treatment after surgery
  Other Names: Chemoradiotherapy

SUMMARY:
SMARCB1-deficient sinonasal carcinoma is very locally advanced malignancy at diagnosis which often precluded upfront radical resection. The investigators are now proposing a phase II single-arm study on tazemetostat in combination with docetaxel, cisplatin and 5-FU (known as TPF regimen) as preoperative therapy for locally advanced non-metastatic SMARCB1 (INI-1)-deficient sinonasal carcinoma, followed by radical resection and/or post-operative radiation therapy (with or without concurrent chemotherapy), and tazemetostat for another 6 months. It is hypothesized that addition of tazemetostat will improve objective response rate, resectability rate, orbit preservation rate after surgery, and hopefully survival outcomes with manageable safety profiles.

DETAILED DESCRIPTION:
SMARCB1 (INI-1)-deficient sinonasal carcinoma is a rare but locally aggressive malignancy of the nasal cavity and paranasal sinuses, representing about only 1 % of all head and neck malignancies. It is characterized by loss of INI-1 in the tumour cells under immunohistochemical staining. The overwhelming majority of INI-1 deficient sinonasal carcinoma presents very late at diagnosis, owing to its very similar clinical presentation to other benign conditions like allergic rhinitis, nasal polyps, chronic sinusitis, and some more common malignancies like human papilloma virus-associated squamous cell carcinoma, extranodal NK/T cells lymphoma, mucosal melanoma. Therefore, complete surgical removal remains very challenging and most of the time impossible.

Currently, aggressive multimodality treatment of INI-1-deficient sinonasal carcinomas is based on experience with other sinonasal malignancies including case series of sinonasal undifferentiated carcinoma. Upfront surgical resection for potentially resectable cases, followed by adjuvant radiation therapy or adjuvant chemoradiation. Also under investigation is the use of induction chemotherapy followed by surgery and adjuvant radiation in the treatment of sinonasal malignancy.

In view of the above, the investigators are now proposing a phase II single-arm study on tazemetostat in combination with TPF as preoperative therapy for locally advanced non-metastatic SMARCB1 (INI-1)-deficient sinonasal carcinoma, followed by radical resection and/or post-operative radiation therapy (with or without concurrent chemotherapy), and tazemetostat for another 6 months. It is hypothesized that addition of tazemetostat will improve objective response rate, resectability rate, orbit preservation rate, and hopefully survival outcomes with manageable safety profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females are >18 years of age with body weight ≥40kg at the time of providing voluntary written informed consent.
2. Voluntarily sign the written informed consent and demonstrated willingness and ability to comply with all aspects of the protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF), and undergoing treatment and scheduled visits and examinations including follow up during the study period,
3. Histologically and/or cytologically confirmed locally advanced (T3-T4bN0-N3M0) non-metastatic SMARCB1 (INI-1)-deficient sinonasal carcinoma
4. For subjects who have experienced any clinically significant toxicity related to a prior anticancer treatment (i.e., chemotherapy, immunotherapy, and/or radiotherapy): at the time the subject provides voluntary written informed consent, all toxicities have either resolved to grade 1 per NCI CTCAE Version 5.0 OR are clinically stable and no longer clinically significant.
5. Have measurable disease as defined by RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Must have a life expectancy of at least 12 weeks before enrollment.
8. Time between prior anticancer therapy and first dose of tazemetostat as follows:

   Cytotoxic chemotherapy - At least 21 days Noncytotoxic chemotherapy (e.g., small molecule inhibitor) - At least 14 days. Nitrosoureas - At least 6 weeks. Monoclonal antibody - At least 28 days.
9. Adequate haematological functions at baseline before commencement of study medication as defined below:

   i. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/liter without growth factor support (filgrastim or pegfilgrastim) for at least 14 days; and ii. Platelets ≥ 100 × 10^9/liter evaluated at least 7 days after platelet transfusion; and iii. Hemoglobin ≥ 9.0 x 10 /litre with blood transfusion allowed before study entry; and after treatment commencement
10. Adequate liver function as defined at baseline before commencement of study medication below:

    Total bilirubin ≤ 1.5 × the upper limit of normal (ULN) (except for unconjugated hyperbilirubinemia of Gilbert's syndrome) Alkaline phosphatase (ALP) (in the absence of bone disease), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN.
11. Adequate renal function as defined below:

    Creatinine < 2.0 or calculated creatinine clearance ≥ 35 mL/minute per the Cockcroft and Gault formula
12. For women of childbearing potential, a negative serum or urine pregnancy test within 14 days prior to the start of treatment. Women will be considered postmenopausal if they are amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    i.) Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy). ii.) Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and partner) to use a highly effective form(s) of contraception that results in a low failure rate (<1% per year) when used consistently and correctly, starting during the screening period, continuing throughout the entire program period, and six months for female and at least three months for male patients after taking the last dose of tazemetostat.

Exclusion Criteria:

1. Pre-existing or co-existing epithelioid sarcoma.
2. Has a prior history of T-Cell lymphoblastic lymphoma, T-cell acute lymphoblastic leukemia, myelodysplastic syndrome, acute myeloid leukemia, or myeloproliferative neoplasm.
3. Have undergone a solid organ transplant.
4. Prior malignancy in the past 5 years.
5. Confirm pregnant or breastfeeding.
6. Prior exposure to tazemetostat or other inhibitor(s) of EZH2.
7. On investigational therapy within 21 days at time of recruitment.
8. Uncontrolled central nervous system (CNS) metastases requiring steroids.
9. On medications that are known potent CYP3A4 inducers/inhibitors (including St. John's wort)
10. Unwilling to exclude Seville oranges, grapefruit juice, and grapefruit from their diet.
11. Had major surgery within 4 weeks before the first dose of study drug. Note: Minor surgery (e.g., minor biopsy of extracranial site, central venous catheter placement, shunt revision) is permitted within 1 week prior to enrollment.
12. Unable to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, vomiting) that might impair the bioavailability of tazemetostat.
13. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II (Appendix 3), uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac ventricular arrhythmia.
14. Have an active infection requiring systemic therapy.
15. Known hypersensitivity to any component of tazemetostat.
16. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the subject's participation in this study OR interfere with their ability to receive study treatment or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Best objective response | 48 months
  Best objective response
R0 resection rate | 48 months
  R0 resection rate

SECONDARY OUTCOMES:
R1 resection rate | 48 months
  R1 resection rate
Complete pathological response rate | 48 months
  Complete pathological response rate
Orbit preservation rate | 48 months
  Orbit preservation rate defined as the rate that sums up that of orbit preservation surgery with a clear resection and that of radical chemoradiation after induction TPF and tazemetostat
Progression-free survival | 48 months
  Progression-free survival
Overall survival | 48 months
  Overall survival
Incidence of treatment-related side effects | 48 months
  Incidence of treatment-related side effects as determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Victor Ho Fun Lee, MD, Principal Investigator — Department of Clinical Oncology, The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.